CLINICAL TRIAL: NCT05608590
Title: Tubal Flushing With Oil-based Contrast During HSG in Subfertile Women: Is Early Flushing Effective and Cost-effective as Compared to Delayed Flushing? - H2Oil-timing Study
Brief Title: What is the Best Moment for Performing an HSG in Women With a Unfulfilled Childwish
Acronym: H2Oil-timing
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Prof. Velja Mijatovic, Professor, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL62838.029.18; 2018.004153.24 (EudraCT Number); NL7926 (Other: NTR)
Record Dates: First submitted 2022-07-18; First posted 2022-11-08 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Female Infertility
Keywords: Infertility; Fallopian tubes; Hysterosalpingography; Tubal flushing; Pregnancy; Live birth; Cost-effectiveness; Randomized controlled trial
MeSH Terms: conditions — Infertility, Female; Infertility | interventions — Ethiodized Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct HSG during fertility work-up (Experimental): Tubal flushing at HSG with Lipiodol® (oil-based contrast medium) (max. 15mL) incorporated in the fertility work-up
  Interventions: Drug: Lipiodol UltraFluid
- Delayed HSG 6 months after completing fertility work-up (Active Comparator): Tubal flushing at HSG with Lipiodol® (oil-based contrast medium) (max. 15mL) after a 6 months waiting period after completion of fertility work-up
  Interventions: Drug: Lipiodol UltraFluid

INTERVENTIONS:
Drug: Lipiodol UltraFluid — The investigational product is an oil-based contrast medium, Lipiodol® (Guerbet). Lipiodol® is a solution of ethyl esters of iodized fatty acids of poppy seed oil equivalent to 480mg I /ml and is a licensed contrast agent in the Netherlands (RVG 02806, see SmPC D2). The maximum amount of Lipiodol® per HSG procedure is 15 ml.
  Other Names: Oil-based contrast

SUMMARY:
The aim of this study is to determine whether direct tubal flushing with oil-based contrast at HSG incorporated in the fertility work-up results in 10% more ongoing pregnancies and a shorter time to pregnancy, which will therefore be effective and cost-effective compared to delayed tubal flushing 6 months after fertility work-up is completed in women at low risk for tubal pathology.

DETAILED DESCRIPTION:
Rationale: The investigators hypothesize that direct tubal flushing with oil-based contrast at HSG incorporated in the fertility work-up results in 10% more ongoing pregnancies and a shorter time to pregnancy compared to delayed tubal flushing 6 months after fertility work-up is completed in women at low risk for tubal pathology, which will lead to a reduction in the need for expensive fertility treatments like IVF and/or ICSI, and will therefore be an effective and cost effective strategy.

Objective: The aim of this study is to determine whether direct tubal flushing with oil-based contrast at HSG incorporated in the fertility work-up results in 10% more ongoing pregnancies and a shorter time to pregnancy, which will therefore be effective and cost-effective compared to delayed tubal flushing 6 months after fertility work-up is completed in women at low risk for tubal pathology.

Study design: The investigators plan a multicentre randomized controlled trial with an economic analysis alongside it. Infertile women at low risk for tubal pathology will be randomized to direct tubal flushing with oil-based contrast incorporated in the fertility work-up or delayed tubal flushing 6 months after fertility work-up is completed.

Study population: Infertile women 18-38 years of age, who have a spontaneous menstrual cycle and at low risk for tubal pathology, undergoing fertility work-up.

Intervention (if applicable): Direct tubal flushing with oil-based contrast at HSG as part of the fertility work-up compared to delayed tubal flushing 6 months after the fertility work-up is completed.

Main study parameters/endpoints: The primary outcome is time to live birth, calculated from positive pregnancy test and within 12 months after randomization.

Our hypothesis is that tubal flushing at HSG with oil-based contrast incorporated in the fertility work-up will result in 10% more ongoing pregnancies and a shorter time to pregnancy, and thus reducing the need for ART and reducing costs.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: As two strategies are compared (tubal flushing with oil-based contrast at HSG incorporated in the fertility work-up versus 6 months after completion of fertility work-up) that are already applied in current practice, no additional risks or burdens are expected from the study.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18-39 years of age
* Spontaneous menstrual cycle
* Perceived low risk for tubal pathology
* Undergoing fertility work-up

Exclusion Criteria:

* Women with known endocrine disorders (e.g. the polycystic ovary syndrome, diabetes, hyperthyroidism and hyperprolactinemia. Except for well managed hypothyroidism with TSH between 0.3 and 2.5mIU/l)
* Ovulation disorders defined as less than eight menstrual cycles per year
* Iodine allergy
* Male subfertility defined as a post-wash total motile sperm count < 1 x10^6 spermatozoa/ml
* Not willing or able to sign the consent form

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 554 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Time to live birth | 6 months
  Calculated from the last menstrual bleeding within 6 months after randomization
Time to live birth | 12 months
  Calculated from the last menstrual bleeding within 12 months after randomization

SECONDARY OUTCOMES:
Number of live births | 6 months
  Defined as the birth of a live born baby, after 24 weeks gestation
Number of live births | 12 months
  Defined as the birth of a live born baby, after 24 weeks gestation
Number of ongoing pregnancies | 6 and 12 months
  Defined as the presence of a heart beat at 10 to 12 weeks gestation
Number of ongoing pregnancies | 6 months
  Defined as the presence of a heart beat at 10 to 12 weeks gestation
Number of clinical pregnancies | 12 months
  Defined as gestational sac detected on ultrasonography
Number of miscarriages | 6 months
  Presence of non-vitality on ultrasound or spontaneous loss of pregnancy
Number of miscarriages | 12 months
  Presence of non-vitality on ultrasound or spontaneous loss of pregnancy
Number of ectopic pregnancies | 6 months
  Embryo implanted outside the uterine cavity
Number of ectopic pregnancies | 12 months
  Embryo implanted outside the uterine cavity
Number of multiple pregnancies | 6 months
  Pregnancy of two or more foetuses
Number of multiple pregnancies | 12 months
  Pregnancy of two or more foetuses
Number of complication after HSG | One month after HSG
  e.g. intravasation or infection
Number of pregnancy complications | 6 months
  e.g. pre-term birth, hypertension
Number of pregnancy complications | 12 months
  e.g. pre-term birth, hypertension
Number of still births | 12 months
  Death or loss of the baby before or during
Number of still births | 6 months
  Death or loss of the baby before or during
Incidence of thyroid dysfunction after HSG | One month after HSG
  TSH and fT4 measurement (blood test)
Number of cycles of artificial reproductive techniques | 6 and 12 months
  Number of cycles of IUI and IVF/ICSI
Number of cycles of artificial reproductive techniques | 6 months
  Number of cycles of IUI and IVF/ICSI
Number of cycles of artificial reproductive techniques | 12 months
  Number of cycles of IUI and IVF/ICSI
Neonatal thyroid dysfunction | Within one week after birth
  Screening on congenital thyroid dysfunction postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No